CLINICAL TRIAL: NCT05869552
Title: Preventing Suicide Among Sexual and Gender Diverse Young Adults in Primary Care: CRT
Brief Title: Preventing Suicide Among Sexual and Gender Diverse Young Adults in Primary Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elizabeth Arnold (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor-Investigator, Elizabeth Arnold, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 86014; SP-2020C3-21020-IC (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Suicide; Suicidal Ideation
Keywords: depression; Self-Injurious Behavior; sexual and gender minority youth
MeSH Terms: conditions — Suicide; Suicidal Ideation; Depression; Self-Injurious Behavior; Coitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suicidal Teens Accessing Treatment - Primary Care (STAT-PC) (Experimental): This group will participate in a brief, suicide prevention intervention based on motivational interviewing that focuses on mental health care seeking behavior, problem-solving, and referrals plus brief case management that has been adapted.
  Interventions: Other: STAT-PC
- Youth-Nominated Support Team (YST-III) (Experimental): This group will participate in a brief, suicide prevention intervention originally developed for youth who have been psychiatrically hospitalized due to a suicide attempt or suicidal ideation that has been adapted.
  Interventions: Other: YST-III

INTERVENTIONS:
Other: STAT-PC — STAT-PC is an adapted version of Suicidal Teens Accessing Treatment after an ED Visit (STAT-ED). It is a brief intervention based on motivational interviewing (MI) that focuses on mental health care seeking behavior, problem-solving, and referrals plus brief case management. The intervention will consist of an initial session with the youth focusing on accessing mental health care plus case management calls. The interventionist will also be available to assist with referrals for connection to other services later during the study period as needed for up to three months. The intervention may include contact with the youth's mental health provider to make sure linkages are made.
  Other Names: Suicidal Teens Accessing Treatment - Primary Care
  Arms: Suicidal Teens Accessing Treatment - Primary Care (STAT-PC)
Other: YST-III — YST-III is an adapted version of Youth-Nominated Support Team for Suicidal Adolescents (YST-II). The intervention is a brief intervention originally developed for youth who have been psychiatrically hospitalized due to a suicide attempt or suicidal ideation (SI). Participants will nominate supportive adults (age 18 and older) from their lives who agree to provide ongoing contact and support for up to 3 months. YST-III will include an introductory session with the youth who will nominate their support persons plus referrals for mental health services. The support persons will receive training and support on how to best support their youth partner and then ongoing calls to support them in working with their youth partner for up to 3 months.
  Other Names: Youth-Nominated Support Team- III
  Arms: Youth-Nominated Support Team (YST-III)

SUMMARY:
The overall aim of this study is to reduce suicide among sexual and gender diverse youth ages 18-24 years old. This study will compare the effectiveness of two brief suicide prevention interventions that have been adapted for use with this population to use in primary care via telehealth and will recruit youth from primary care clinics in multiple metropolitan areas. The primary study outcome is suicidal ideation. Each clinic will be randomly assigned to deliver one of the two study interventions.

ELIGIBILITY:
Inclusion Criteria:

* be aged 18-24 at the time of enrollment
* not have received mental health services in the past 90 days, excluding medication and case management
* English-speaking
* screen positive for suicide risk

Exclusion Criteria:

* are actively suicidal
* have a developmental disability that would preclude them from participating in the study intervention
* who are impaired due to psychosis, mania, or substance use that would prevent them from providing consent.
* Participants will also be excluded at YST-III sites if they are unable to identify a minimum of one support person to participate in the intervention with them

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — To enroll, participants must identify as a sexual or gender minority individual (i.e., LGBTQ+) and be a patient of the one the clinic sites
Enrollment: 1485 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change in suicidal ideation as measured by the Adult Suicidal Ideation Questionnaire (ASIQ) | baseline and months 1, 3, 6
  ASIQ is a 25-item, self-report assessment of suicidal thoughts designed specifically for adult populations. Possible scores range from 1 (Not at All) to 6 (Extreme), with lower scores indicating less severe suicidal ideation (better outcome).

SECONDARY OUTCOMES:
Change in number of mental healthcare service utilization as measured by Emergency Department Screen for Teens at Risk for Suicide (ED-STARS) mental health service utilization check list | baseline and months 1, 3, 6
  ED-STARS mental health service utilization check list will be used to assess the number of different types of mental health services that participants receive
Change in number of suicide attempts | baseline and months 1, 3, 6
  measured by the number of suicide attempts using the Columbia-Suicide Severity Rating Scale (CSSRS)
Deaths by suicide | baseline to 6 months
  The data on any reported deaths due to suicide during the study period will be collected.
Change in depressive symptoms as measured by Center for Epidemiologic Studies Depression Scale-Revised CESD-R | baseline and months 1, 3, 6
  CESD-R is a 20-item measure of depression that assesses the duration symptoms across a period of two weeks. Possible scores range from 0-60, with lower scores indicating less depressive symptoms (better outcome).
Change in social support as measured by the Multidimensional Scale of Perceived Social Support (MSPSS) | baseline and months 1, 3, 6
  12-item measure with three subscales that assesses family, friend, and significant other support. Response categories are on a 7-point Likert-scale from 1=very strongly disagree to 7=very strongly agree. The overall score will be used to assess change. The 12-item MSPSS scale has a mean continuous score ranging from 1-84. Higher scores indicate greater perceived social support (better outcome).
Change in internalized stigma as measured by Internalized Transphobia Scale (ITS)-adapted | baseline and months 1, 3, 6
  an adapted version of the Internalized Transphobia Scale (ITS). The measure consists of 22 questions. Possible score ranges from 1-4 with lower scores indicating less internalized stigma (better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Arnold, PhD, Principal Investigator — University of Kentucky
Locations (3):
- United States (3):
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Steve Hicks School of Social Work at the University of Texas at Austin, Austin, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be deposited in the Patient-Centered Outcomes Data Repository as required by the funder.
Supporting Information: Study Protocol
Time Frame: By the date that the Final Research Report is accepted by the funder
Access Criteria: Researchers must go through the Patient-Centered Outcomes Data Repository to request access to the de-identified data through their process.